CLINICAL TRIAL: NCT06187298
Title: The Adjuvant Synergistic Therapeutic Effect of Oral Berberine and Curcumin Alleviates Symptoms of Irritable Bowel Syndrome: Results From a Real-life Setting Clinical Intervention Study
Brief Title: Effect of Oral Combined Berberine and Curcumin Pharmacological Therapy on IBS
Status: Completed | Type: Observational
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Other Study IDs: LUMHS/UOL-BE/16.12.2023
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Curcumin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: A combined supplement of Berberine and Curcumin (Enterophytol® PLUS) alongside standard of care — (Enterophytol® PLUS) alongside standard of care

SUMMARY:
Irritable bowel syndrome (IBS) is a prevalent, chronic functional gastrointestinal (GI) disorder, characterized by recurrent abdominal discomfort (pain) associated with altered bowel movements. IBS has a considerable negative impact on people's quality of life (QoL). There is currently no specific treatment available for IBS; most of the therapeutic management is symptomatic. Reported evidence suggest that BBR and CUR can alleviate symptoms of IBS through their multiple pharmacological effects including preventing stress-induced intestinal inflammation and visceral hypersensitivity, reducing bowel motility, and regulating intestinal permeability, gut microme and gut-brain axis.

DETAILED DESCRIPTION:
Aim of the study:

The present clinical study aimed to assess the synergestic therapeutic effect of a combined supplement of standardised extract of BBR and CUR (Enterophytol® PLUS, 200 mg BBR, 49 mg CUR) in the management of IBS.

Method : This was an in real-life setting pragmatic, observational, retrospective, non-controlled and non-randomized clinical trial involving 146 patients with IBS, enrolled in General Practitioner clinics and Pharmacies in Belgium from Aug 2020 to May 2022. The supplement was used as two tablets daily for 2-months, alongside routine IBS care.

ELIGIBILITY:
Inclusion Criteria:

* Self-completion of simplified form of the Rome IV IBS diagnostic criteria
* Had IBS symptoms that appeared before the age of 50
* Used Enterophytol® PLUS as complementary therapy as two tablets a day for 2-months

Exclusion Criteria:

* Those with involuntary weight loss
* Family history of chronic inflammatory bowel disease, colorectal cancer, celiac disease, rectal discharge, nocturnal symptoms, fever, and abnormalities on clinical examination (abdominal mass, signs of anaemia).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients enrolled at GP clinics and Pharmacies in Belgium
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in the overall IBS Severity Index | At 2 months
  Reduction in the IBS overall symptoms severity index

SECONDARY OUTCOMES:
Change in weekly frequency of stool passage | At 2 months
  Treatment effect on patient's weekly stool passage frequency
Change in the stool form | At 2 months
  Change in the physical appearance of patient's stool
Change in the number of IBS standard of care drugs | At 2 months
  Treatment effect on patient's need for IBS drugs
Number of patients with side effects | At 2 months
  Treatment safety and tolerability
Number of patients with treatment satisfaction | At 2 months
  Treatment satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University of Medical and Health Sciences, Jāmshoro, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michel P H, Ahn SA, Rousseau MF, Seidel L, Albert A, Janssens I, Dierckxsens Y, Khan A. Potential synergistic antihyperglycemic effects of co-supplemental Amla and Olive extracts in hyperlipidemic adults with prediabetes and type 2 diabetes: results from a real-life clinical study. Front Nutr. 2024 Oct 3;11:1462292. doi: 10.3389/fnut.2024.1462292. eCollection 2024. PMID 39421612